CLINICAL TRIAL: NCT01803230
Title: Effects of Creatine Supplementation on Cognitive Function in Children
Brief Title: Creatine Supplementation on Cognition in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Creatine in Children
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: children
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo (dextrose)
  Interventions: Dietary Supplement: Placebo
- creatine (Experimental): creatine supplementation
  Interventions: Dietary Supplement: creatine supplementation

INTERVENTIONS:
Dietary Supplement: creatine supplementation — creatine supplementation
  Arms: creatine
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
Creatine supplementation may improve cognitive function in elderly and vegetarian individuals. This study aims to investigate the role of creatine supplementation on cognitive function in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* healthy children
* age between 10 to 12 years of age

Exclusion Criteria:

* cognitive impairment
* vegetarian diet
* use of creatine in the past 6 months
* chronic kidney disease

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
cognitive function | 7 days
  assessed by a battery of cognitive tests as follows: colors and words attention test, controlled words association test, memory and figures learning, mental flexibility test and inhibitory control, digit span test, and intelligence quotient.

SECONDARY OUTCOMES:
tissue creatine content | 7 days
  as assessed by 1H-MRS.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil